CLINICAL TRIAL: NCT01986478
Title: Topcon 3D OCT-1 Maestro and 3D OCT-2000 Optical Coherence Tomography Systems: Reference Database Study
Brief Title: OCT Reference Database
Status: Completed | Type: Observational
Sponsor: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Organization: Topcon Corporation (Industry)
Other Study IDs: DC-001
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normal: Normal results from clinical exam and free of ocular pathology

SUMMARY:
To collect data for a reference database.

DETAILED DESCRIPTION:
Collection of multiple subjects to create a reference database.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 years of age or older on the date of informed consent
2. Subjects able to understand the written informed consent and willing to participate as evidenced by signing the informed consent
3. Subjects presenting at the site with normal eyes (eyes without pathology)
4. IOP ≤ 21 mmHg bilaterally
5. BCVA 20/40 or better (each eye)
6. Both eyes must be free of eye disease

Exclusion Criteria:

1. Subjects unable to tolerate ophthalmic imaging
2. Subject with ocular media not sufficiently clear to obtain acceptable OCT images
3. HFA visual field (24-2 Sita Standard, white on white) result abnormal, defined as GHT 'Outside Normal Limits' and/or PSD < 5%
4. HFA visual field (24-2 Sita Standard, white on white) result unreliable (based on manufacturer's recommendation), defined as fixation losses > 33% or false positives > 25%, or false negatives > 25%
5. Presence of any ocular pathology except for cataract
6. Previous ocular surgery or laser treatment, other than uncomplicated refractive procedure or cataract surgery, performed within six months prior to study scanning
7. Narrow angle
8. History of leukemia, dementia or multiple sclerosis
9. Concomitant use of hydroxychloroquine and chloroquine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects that are Normal
Sampling Method: Non-Probability Sample
Enrollment: 389 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Retinal Thickness | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sinai, PhD, Principal Investigator — Senior Manager Product Planning Group
Locations (5):
- United States (5):
  - Horizon Eye Specialist & Laser Center, Scottsdale, Arizona
  - Valley Eyecare Center, Livermore, California
  - Keck School of Medicine, Los Angeles, California
  - Western University of Health Sciences, Pomona, California
  - Stat University of New York College of Optometry, New York, New York